CLINICAL TRIAL: NCT06790836
Title: Correlation of Fractional Flow Reserve Computed Tomography (FFR CT) Findings With Invasive FFR in Coronary Artery Disease (CAD) in a Multi-ethnic Cohort- a Retrospective Study
Brief Title: Correlation of FFR CT With Invasive FFR in Multi-ethnic Cohort- a Retrospective Study
Status: Not yet recruiting | Type: Observational
Sponsor: Sandwell & West Birmingham Hospitals NHS Trust (Other)
Collaborators: Aston University (Other)
Responsible Party: Principal Investigator, Vinoda Sharma, Chief Investigator, Sandwell & West Birmingham Hospitals NHS Trust
Other Study IDs: IRAS #339186
Record Dates: First submitted 2025-01-18; First posted 2025-01-24 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2025-01

CONDITIONS: Coronary Artery Disease
Keywords: FFR CT; Invasive FFR; Comparison
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims to examine the correlation between Fractional Flow Reserve (FFR) FFR Computed Tomography (CT) and invasive FFR in a real-world setting using retrospective analysis of existing data, providing practical insights directly applicable to patient care. By confirming or examining the accuracy of FFR CT in a clinical setting, our analysis could support its broader adoption as a routine non-invasive diagnostic tool potentially (a) reducing the need for invasive testing (b) minimising associated risks, and(c) lowering healthcare costs and provide fresh insights into non-invasive coronary diagnostics. Our findings will also help understand the relevance of these tests across different ethnic groups and the population we serve.

DETAILED DESCRIPTION:
This retrospective study will analyse the existing Computed Tomography Coronary Angiogram (CTCA) database for patients treated at Sandwell and West Birmingham (SWBH) National Health Service (NHS) Trust between January 1, 2019, and December 31, 2023, with the clinical team screening the database to identify patients who fit with the eligibility criteria.

The proposed study is a retrospective analysis of the clinical and imaging data over a five-year period in patients with stable chest pain (approximately 500 patients), who underwent CTCA, FFR CT, and invasive FFR at SWBH NHS Trust. The study will assess the correlation between these diagnostic measures. The aim of this investigation is to address the ongoing discrepancies in the diagnostic accuracy of FFR CT compared to the gold standard invasive FFR, which persist despite the increasing adoption of FFR CT in clinical practice. While initial trials indicated promising sensitivity and specificity for FFR CT, recent observational studies including one involving 2,298 patients who underwent FFR CT, reported varying positive and negative predictive values, with a low positive predictive value of 49% (24). This variability raised concerns about the reliability of FFR CT across different patient populations, and the real-world accuracy and cost-effectiveness of FFR CT remain subjects of ongoing debate.

This study aims to examine the correlation between FFR CT and invasive FFR in a real-world setting using existing data, providing practical insights directly applicable to patient care. By confirming or examining the accuracy of FFR CT in a clinical setting, our analysis could support its broader adoption as a routine non-invasive diagnostic tool potentially (a) reducing the need for invasive testing (b) minimising associated risks, and(c) lowering healthcare costs and provide fresh insights into non-invasive coronary diagnostics. Our findings will also help understand the relevance of these tests across different ethnic groups and the population we serve.

The patient data will be identified by accessing the CTCA database, and the study will adhere to the STrengthening the Reporting of OBservational studies in Epidemiology (STROBE) guidelines (25).

The eligibility criteria are as follows:

* Patients aged 18 years and above.
* Patients presenting to the hospital with stable chest pain.
* Patients who have undergone both FFR CT and invasive FFR. Ethical approval will be obtained through the Integrated Research Application System (IRAS).

The patient's information will be collected by members of the research team, including demographic data such as age, gender, body mass index (BMI), and cardiovascular risk factors (e.g., smoking, hypertension, and diabetes). Vessel characteristics, including the coronary artery involved, location, and degree of stenosis, will also be recorded. Results of FFR CT and Invasive Coronary Angiogram (ICA) findings (if performed), as well as diagnostic performance metrics-sensitivity, specificity, positive predictive value (PPV), negative predictive value (NPV), and accuracy of FFR CT in comparison to invasive FFR-along with downstream testing and imaging data, will be extracted from the CTCA database. All data will be coded and anonymised to ensure patient confidentiality and stored on NHS Trust computers with individual, password-protected logins. Only members of the research team involved in the study will have access to these computers.

We will ensure all data collected, stored, and used complies with data protection laws, including the General Data Protection Regulation (GDPR) and the UK Data Protection Act 2018. Patient information will be anonymised to maintain confidentiality. The data will be securely stored on NHS computers at SWBH and used solely for this research.

An overview of the patient cohort will be provided, including demographics and clinical characteristics. Additionally, a detailed comparison of the diagnostic accuracy of FFR CT versus invasive FFR will be presented, including sensitivity, specificity, PPV, NPV, and overall accuracy.

Furthermore, the correlation between FFR CT and invasive FFR values will be explored, with a focus on any significant findings or discrepancies that may arise, offering insights into the diagnostic performance of FFR CT in comparison to the gold standard.

Statistical analysis will be performed using SPSS software, version 27. Continuous variables will be presented as mean ± standard deviation (SD) and compared using the Mann-Whitney U test or Analysis of Variance (ANOVA), as appropriate. Categorical variables will be expressed as percentages and compared using the chi-square test. Sensitivity, specificity, PPV, and NPV will be calculated based on the correlation between FFR CT and invasive FFR.

Inclusion Criteria:

Patients meeting all the below criteria will be included.

•≥18 years

* Stable •patients with suspected CAD
* Patients who underwent CTCA, FFR CT and had an invasive FFR.
* CTCA images of high-quality for analysis, with clear visualisation of coronary arteries and minimal artifacts.

Exclusion criteria:

Patients meeting any of the following criteria will be excluded.

* <18 years of age
* Did not undergo FFR CT
* Inadequate quality/degraded CTCA images Online database on password protected NHS TRUST computer to collect demographic parameters of all patients i.e. age, sex, BMI along with history of disease, coexisting morbidities like hypertension, diabetes and hyperlipidaemia procedural and outcome information.

Demographics (age, gender, ethnicity socio economic status), BMI and cardiovascular risk factors) vessel characteristics, FFR CT values and invasive FFR values will be obtained.

Categorical variables will be compared by chi square test or Fisher's test and continuous variables will be compared by Mann Whitney U test Ethical approval for this retrospective study will be obtained through IRAS application.

References

1. Organization WH. Cardiovascular diseases (CVDs) 2021 [Available from: https://www.who.int/news-room/fact-sheets/detail/cardiovascular-diseases-(cvds).
2. Writing Group M, Mozaffarian D, Benjamin EJ, Go AS, Arnett DK, Blaha MJ, et al. Heart Disease and Stroke Statistics-2016 Update: A Report From the American Heart Association. Circulation. 2016;133(4):e38-360.
3. Yamagishi M, Tamaki N, Akasaka T, Ikeda T, Ueshima K, Uemura S, et al. JCS 2018 Guideline on Diagnosis of Chronic Coronary Heart Diseases. Circulation Journal. 2021;85(4):402-572.
4. Wolk MJ, Bailey SR, Doherty JU, Douglas PS, Hendel RC, Kramer CM, et al. ACCF/AHA/ASE/ASNC/HFSA/HRS/SCAI/SCCT/SCMR/STS 2013 multimodality appropriate use criteria for the detection and risk assessment of stable ischemic heart disease: a report of the American College of Cardiology Foundation Appropriate Use Criteria Task Force, American Heart Association, American Society of Echocardiography, American Society of Nuclear Cardiology, Heart Failure Society of America, Heart Rhythm Society, Society for Cardiovascular Angiography and Interventions, Society of Cardiovascular Computed Tomography, Society for Cardiovascular Magnetic Resonance, and Society of Thoracic Surgeons. J Am Coll Cardiol. 2014;63(4):380-406.
5. Douglas PS, Hoffmann U, Lee KL, Mark DB, Al-Khalidi HR, Anstrom K, et al. PROspective Multicenter Imaging Study for Evaluation of chest pain: rationale and design of the PROMISE trial. American heart journal. 2014;167(6):796-803. e1.
6. CT coronary angiography in patients with suspected angina due to coronary heart disease (SCOT-HEART): an open-label, parallel-group, multicentre trial. The Lancet. 2015;385(9985):2383-91.
7. Alfakih K, Byrne J, Monaghan M. CT coronary angiography: a paradigm shift for functional imaging tests. Open Heart. 2018;5(1):e000754.
8. (NICE) NIfHaCE. HeartFlow FFRCT for estimating fractional flow reserve from coronary CT angiography. 2017.
9. Cremer PC, Nissen SE. The National Institute for Health and Care Excellence update for stable chest pain: poorly reasoned and risky for patients. Heart. 2017;103(13):972-4.
10. Pijls NHJ, De Bruyne B, Peels K, Van Der Voort PH, Bonnier HJRM, Bartunek J, et al. Measurement of Fractional Flow Reserve to Assess the Functional Severity of Coronary-Artery Stenoses. New England Journal of Medicine. 1996;334(26):1703-8.
11. Achenbach S, Rudolph T, Rieber J, Eggebrecht H, Richardt G, Schmitz T, et al. Performing and interpreting fractional flow reserve measurements in clinical practice: an expert consensus document. Interventional Cardiology Review. 2017;12(2):97.
12. Xaplanteris P, Fournier S, Pijls NHJ, Fearon WF, Barbato E, Tonino PAL, et al. Five-Year Outcomes with PCI Guided by Fractional Flow Reserve. New England Journal of Medicine. 2018;379(3):250-9.
13. De Bruyne B, Pijls NHJ, Kalesan B, Barbato E, Tonino PAL, Piroth Z, et al. Fractional Flow Reserve-Guided PCI versus Medical Therapy in Stable Coronary Disease. New England Journal of Medicine. 2012;367(11):991-1001.
14. Scoccia A, Tomaniak M, Neleman T, Groenland FTW, Plantes ACZD, Daemen J. Angiography-Based Fractional Flow Reserve: State of the Art. Current Cardiology Reports. 2022;24(6):667-78.
15. Members TF, Montalescot G, Sechtem U, Achenbach S, Andreotti F, Arden C, et al. 2013 ESC guidelines on the management of stable coronary artery disease: The Task Force on the management of stable coronary artery disease of the European Society of Cardiology. European Heart Journal. 2013;34(38):2949-3003.
16. Kurata A, Fukuyama N, Hirai K, Kawaguchi N, Tanabe Y, Okayama H, et al. On-Site Computed Tomography-Derived Fractional Flow Reserve Using a Machine-Learning Algorithm - Clinical Effectiveness in a Retrospective Multicenter Cohort -. Circulation Journal. 2019;83(7):1563-71.
17. Kimura T, Shiomi H, Kuribayashi S, Isshiki T, Kanazawa S, Ito H, et al. Cost analysis of non-invasive fractional flow reserve derived from coronary computed tomographic angiography in Japan. Cardiovascular Intervention and Therapeutics. 2015;30(1):38-44.
18. Nørgaard BL, Leipsic J, Gaur S, Seneviratne S, Ko BS, Ito H, et al. Diagnostic performance of noninvasive fractional flow reserve derived from coronary computed tomography angiography in suspected coronary artery disease: the NXT trial (Analysis of Coronary Blood Flow Using CT Angiography: Next Steps). J Am Coll Cardiol. 2014;63(12):1145-55.
19. Koo BK, Erglis A, Doh JH, Daniels DV, Jegere S, Kim HS, et al. Diagnosis of ischemia-causing coronary stenoses by noninvasive fractional flow reserve computed from coronary computed tomographic angiograms. Results from the prospective multicenter DISCOVER-FLOW (Diagnosis of Ischemia-Causing Stenoses Obtained Via Noninvasive Fractional Flow Reserve) study. J Am Coll Cardiol. 2011;58(19):1989-97.
20. Gray AJ, Roobottom C, Smith JE, Goodacre S, Oatey K, O'Brien R, et al. Early computed tomography coronary angiography in patients with suspected acute coronary syndrome: randomised controlled trial. BMJ. 2021:n2106.
21. Curzen N, Nicholas Z, Stuart B, Wilding S, Hill K, Shambrook J, et al. Fractional flow reserve derived from computed tomography coronary angiography in the assessment and management of stable chest pain: the FORECAST randomized trial. European Heart Journal. 2021;42(37):3844-52.
22. Upadhyaya SGN, Santhirasekaram A, Dharas M, Yousif A, D'sa A, Das I, et al. OSCRIS; An Efficient and Patient preferred Cardiac CT service. Journal of Cardiovascular Computed Tomography. 2019;13(1):S9.
23. (NHS) NHS. Innovation and Technology Payment. (2018-2021).
24. Mittal TK, Hothi SS, Venugopal V, Taleyratne J, O'Brien D, Adnan K, et al. The Use and Efficacy of FFR-CT. JACC: Cardiovascular Imaging. 2023;16(8):1056-65.
25. Von Elm E, Altman DG, Egger M, Pocock SJ, Gøtzsche PC, Vandenbroucke JP. The Strengthening the Reporting of Observational Studies in Epidemiology (STROBE) statement: guidelines for reporting observational studies. Journal of Clinical Epidemiology. 2008;61(4):344-9.

ELIGIBILITY:
Inclusion Criteria:

* •≥18 years

  * Stable •patients with suspected CAD
  * Patients who underwent CTCA, FFR CT and had an invasive FFR.
  * CTCA images of high-quality for analysis, with clear visualisation of coronary arteries and minimal artifacts.

Exclusion Criteria:

* •<18 years of age

  * Did not undergo FFR CT
  * Inadequate quality/degraded CTCA images

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The existing CTCA database for patients treated at Sandwell and West Birmingham NHS Trust between January 1, 2019, and December 31, 2023, with the clinical team screening the database to identify patients who fit with the eligibility criteria.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Correlation between FFR CT and invasive FFR. | 6 months
  Correlation as mesured by positive predicitve value, negative predictive value, sensitivity and specificity

SECONDARY OUTCOMES:
Assess the downstream testing after FFR CT | 6 months
  By assessing the rates and results of invasive coronary angiography

CONTACTS AND LOCATIONS:
Locations (1):
- Sandwell and West Birmingham NHS Trust, Birmingham, West Midlands, United Kingdom

IPD SHARING:
Plan to Share IPD: No
This study involves a retrospective database analysis- on completion of analysis and write up, data can be shared on request